CLINICAL TRIAL: NCT04227548
Title: Reference Values for the Ratio of Compound Muscle Action Potential Amplitude Obtained by Nerve Stimulation to That Obtained by Direct Muscle Stimulation
Brief Title: Reference Values for Compound Muscle Action Potential Amplitude Obtained by Direct Muscle Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halit Fidancı, Medical Doctor, Neurology and Clinical Neurophysiology, Adana City Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 30/401
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Critical Illness Polyneuromyopathy
Keywords: Critical illness myopathy; Critical illness neuropathy; direct muscle stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy individuals (Experimental)
  Interventions: Diagnostic Test: needle electromyography

INTERVENTIONS:
Diagnostic Test: needle electromyography — Direct muscle stimulation was performed to deltoid and tibialis anterior muscles with a monopolar needle electrode. Recording was made with a concentric needle electrode.

SUMMARY:
Direct muscle stimulation (DMS) method is one of the electrodiagnostic methods used in the diagnosis of critical illness myopathy (CIM) and critical illness neuropathy (CIN). The ratio of amplitude of compound muscle action potential (CMAP) obtained by nerve stimulation (nCMAP) to amplitude of CMAP obtained by DMS (dmCMAP) can be used to differentiate these two diseases. Although not certain, if the ratio is < 0.5, the diagnosis is thought to be consistent with CIN. The ratio > 0.5 is considered to be a finding supporting CIM. The investigators aimed to find the reference values of the ratio from healthy individuals. A monopolar needle electrode was used for DMS. The dmCMAP and nCMAP were recorded with a concentric needle. The ratio was calculated by using amplitudes of dmCMAP and nCMAP obtained from deltoid and tibialis anterior muscles.

DETAILED DESCRIPTION:
Age, gender, height, weight, body mass index and neurological examination findings of the participants were recorded. Healthy participants were not included if they had; polyneuropathy or a disease such as diabetes mellitus that causes polyneuropathy, complaints such as weakness or paresthesia, a neurodegenerative disease, abnormal neurological examination, myopathy or hereditary polyneuropathy in family history. In addition, healthy participants were excluded if the conventional nerve conduction study and needle electromyography (EMG) findings were abnormal. Median, ulnar, posterior tibial, peroneal, superficial peroneal, sural nerve conduction studies were performed to all participants. Needle EMG and direct muscle stimulation were applied to the deltoid and tibialis anterior muscles of the healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Polyneuropathy
* a disease such as diabetes mellitus that causes polyneuropathy
* complaints such as weakness or paresthesia
* a neurodegenerative disease
* abnormal neurological examination

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the Ratio of Compound Muscle Action Potential Amplitude Obtained by Nerve Stimulation to That Obtained by Direct Muscle Stimulation | 1 hour
  The normal limits of the ratio were the primary outcome criteria. This ratio is high in critical illness myopathy or healthy individuals, while low in ciritical illness neuropathy of broken disease occurs. Considering the study of Lefaucheur et al., at least 23 healthy individuals should be included in the study.(Lefaucheur JP, Nordine T, Rodriguez P, Brochard L (2006) Origin of ICU acquired paresis determined by direct muscle stimulation. J Neurol Neurosurg Psychiatry 77:500-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided